CLINICAL TRIAL: NCT05890118
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics (PK) of RT-111- RaniPill Capsule Containing Ustekinumab - Administered Orally to Healthy Volunteers
Brief Title: Study Evaluating PK of Ustekinumab Administered Orally Via RaniPill™ Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RANI Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT-111-001
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SC Group (Active Comparator): In up to 15 volunteers, 0.5mg of Stelara will be administered subcutaneously and serial blood samples will be collected for PK analysis.
  Interventions: Drug: Stelara
- RT-111 Group 1 (Experimental): In up to 20 volunteers, a RaniPill capsule containing 0.5mg of ustekinumab will be administered and serial blood samples will be collected for PK analysis.
  Interventions: Combination Product: RT-111 (0.5mg)
- RT-111 Group 2 (Experimental): In up to 20 volunteers, a RaniPill capsule containing 0.75mg of ustekinumab will be administered and serial blood samples will be collected for PK analysis.
  Interventions: Combination Product: RT-111 (0.75mg)

INTERVENTIONS:
Drug: Stelara — A commercial formulation of ustekinumab for SC control (0.5mg)
  Arms: SC Group
Combination Product: RT-111 (0.5mg) — RaniPill capsule containing ustekinumab with a dose of 0.5mg
  Arms: RT-111 Group 1
Combination Product: RT-111 (0.75mg) — RaniPill capsule containing ustekinumab with a dose of 0.75mg
  Arms: RT-111 Group 2

SUMMARY:
A prospective, single-center, open-label, phase 1 study evaluating the pharmacokinetics (PK) of ustekinumab administered via the RaniPill™ capsule ("RT-111").

DETAILED DESCRIPTION:
The RaniPill device is a capsule-like ingestible device, which injects a microneedle containing a micro tablet (payload/drug) into the intestinal wall. This is a single-center, prospective, open-label, phase 1 study.

Healthy Volunteers, 18-65 years of age, of any race, recruited from the general population and assigned to one of the following groups:

* Group 1 (SC Control): Stelara®, 0.5mg via SC injection (N= up to 15)
* Group 2: RT-111-0.50 mg (N= up to 20)
* Group 3: RT-111-0.75 mg (N=up to 20)

ELIGIBILITY:
Inclusion Criteria:

1. Participant is ambulatory and between 18 to 65 years of age
2. Body mass index between 19- 32 kg/m2
3. RT-111 ONLY: Female volunteers must be non-menstruating at dosing
4. Female volunteers must be non-pregnant or non-lactating during study participation
5. Male volunteers must agree to use acceptable forms of contraception, if necessary, and to not donate sperm during study participation.
6. Have suitable venous access for blood sampling.
7. In good general health confirmed by medical history, physical examination, and absence of clinically important laboratory abnormalities per Investigator's judgment
8. Participant understands the nature of the study, is willing to comply with protocol defined evaluations, and provide written informed consent

Exclusion Criteria:

1. History of intolerance to Stelara® or its constituents
2. Have a known history of previous exposure to IL-12 and/or IL-23 inhibitors.
3. History (≤10 years) or presence of disease determined by the PI to be clinically significant including:

   1. gastrointestinal (including diverticulitis, stomach ulcers, inflammatory intestinal disease, gastrointestinal perforations/fistulae/intra-abdominal abscess).
   2. any other internal, non-gastrointestinal fistulae that is at an increased risk of bleeding.
   3. hematological (including pancytopenia, aplastic anemia, or blood dyscrasia).
   4. renal, endocrine, hepatic, pulmonary (childhood asthma is allowed), neurologic, psychiatric, metabolic (including known diabetes mellitus), or
   5. allergic disease excluding mild asymptomatic seasonal and food allergies.
4. Have a history of prolonged immunosuppressant therapy or photochemotherapy treatment.
5. Presence or evidence of recent sunburn, scar tissue, tattoo (more than 25% of body area), open sore or branding that, in the opinion of the Investigator, would interfere with interpretation of skin adverse reactions.
6. Have a history of and/or current cardiac disease defined as one of the following:

   1. History of congestive heart failure; angina pectoris requiring anti-anginal medication.
   2. Evidence of transmural infarction on ECG.
   3. History of sustained hypertension (systolic > 180 mmHg and/or diastolic > 100 mmHg), hypertensive crisis or hypertension encephalopathy.
   4. Clinically significant valvular heart disease or severe arterial thromboembolic events.
7. Have a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus, human immunodeficiency virus (HIV) or history of active, latent, or inadequately treated tuberculosis (TB) infection
8. Positive serum pregnancy test for women of childbearing potential at the Screening visit or positive urine pregnancy test with confirmatory serum pregnancy test prior to dosing.
9. Females who are breastfeeding.
10. Have a history of cancer including lymphoma, leukemia, and skin cancer (volunteers with a maximum of 3 surgically resected basal cell carcinoma or squamous cell carcinoma are permitted).
11. Have an illness within 30 days prior to screening, or prior to dosing, that has not resolved and is classed as clinically significant by the Investigator.
12. Any current active infections, including localized infections, or any recent history (within 1 week prior to study drug administration) of active infections (including severe acute respiratory syndrome coronavirus 2 [SARS-CoV-2] based on a positive COVID-19 polymerase chain reaction [PCR] nasopharyngeal swab test), cough or fever, or a history of recurrent or chronic infections.
13. Have had major surgery within 30 days prior to screening or will have an operation between screening and the end of study visit, or have any unhealed wound, including wound dehiscence and wound healing complications requiring medical intervention.
14. Have received live vaccines during the past 4 weeks before Screening or have the intention to receive vaccination during the study period or within 13 weeks after dosing.
15. Have received a Bacillus Calmette-Guerin (BCG) vaccination within 1 year prior to dose administration or is planning to receive a BCG vaccination within 1 year following dose administration.
16. History of alcohol abuse (defined as more than 12 standard drinks per week or more than 4 standard drinks on > 3 days per week; where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]) within 12 weeks prior to the screening visit.
17. Positive drug or alcohol test results. In the event the urinary drug test is positive, the test may be repeated once (at the discretion of the PI) to confirm eligibility.
18. Donation of more than 500 mL of blood within 4 weeks prior to drug administration.
19. Abnormal or irregular bowel movements, in the opinion of the Investigator.
20. Any history of non-traumatic hemorrhage (i.e., any hemorrhage requiring medical intervention) or any condition which may increase bleeding risk including clotting disorders, thrombocytopenia (platelet count < 150,000 per μL) or an international normalized ratio higher than 1.5.
21. Impaired liver function as determined by a serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)> 1.5 x upper limit of normal (ULN). Participants with values between ULN and 1.5 x ULN may be included in the study if considered not clinically significant by the Investigator.
22. Treatment with non-topical medications (including over-the-counter [OTC] medications and herbal remedies such as St. John's Wort extract) within 7 days or 5 half-lives of the drug (whichever is longer) prior to CTM administration, with the exception of multivitamins, vitamin C, food supplements and a limited amount of acetaminophen (up to 2 g in 24 hours, but <1 g in 4 hours) or ibuprofen (<1.2 g per day), which may be used throughout the study.
23. Participants on a higher than the lowest approved therapeutic dose regimen of proton pump inhibitors (see Section 9.1.6 for details)
24. Participants on a H2 receptor antagonists (e.g., famotidine, cimetidine)
25. Consumption of any foods containing poppy seeds within 48 hours prior to screening and admission to the clinical center.
26. Presence of proteinuria (other than trace amounts i.e., +, ++/+++).
27. Personal history of venous thromboembolic events or idiopathic venous thromboembolic events in a first degree relative.
28. Excessive smoking habit (more than 5 cigarettes/day) or drug consumption
29. Other clinically relevant findings per physical or laboratory examination or symptoms of a clinically relevant illness 3 weeks prior to the dose of study drug.
30. Participation in a clinical study with an IP dosing within 60 days or 5 half-lives of that IP (if known), whichever is longer, prior to IP administration in the current study.
31. History which, in the investigator's judgement, makes the participant ineligible or exposes the participant to unacceptable risks
32. Low likelihood, in the Investigator's judgment, to complete the study as required per study plan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Evaluate Cmax of ustekinumab administered via the RaniPill capsule | Within 60 days after ingesting the device
  To obtain PK profiles of single doses of ustekinumab given via RaniPill™ capsule in healthy volunteers over a dose range of 0.5 to 0.75mg. Cmax of ustekinumab will be calculated from the PK profiles.
Evaluate Tmax of ustekinumab administered via the RaniPill capsule | Within 60 days after ingesting the device
  To obtain PK profiles of single doses of ustekinumab given via RaniPill™ capsule in healthy volunteers over a dose range of 0.5 to 0.75mg. Cmax of ustekinumab will be calculated from the PK profiles.
Evaluate AUC of ustekinumab administered via the RaniPill capsule | Within 60 days after ingesting the device
  To obtain PK profiles of single doses of ustekinumab given via RaniPill™ capsule in healthy volunteers over a dose range of 0.5 to 0.75mg. Cmax of ustekinumab will be calculated from the PK profiles.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability of RT-111) | Within 60 days after ingesting the device
  Monitoring and recording of adverse events possibly related to RT-111.

CONTACTS AND LOCATIONS:
Overall Officials: Arvinder Dhalla, PhD, Study Director — RANI Therapeutics
Locations (1):
- Nucleus Network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No